CLINICAL TRIAL: NCT00089765
Title: Pilot Study of Intravitreal Injection of Ranibizumab (rhuFAB V2) for Advanced Ocular Disease of Von Hippel-Lindau (VHL) Disease
Brief Title: Ranibizumab Injections to Treat Retinal Tumors in Patients With Von Hippel-Lindau Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040240; 04-EI-0240
Record Dates: First submitted 2004-08-12; First posted 2004-08-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-08-15

CONDITIONS: Von Hippel-Lindau Syndrome
Keywords: Retinal Angioma; Tumor; Anti-VEGF; Monoclonal Antibody; Macular Edema; Von Hippel-Lindau Disease; VEGF; Ranibizumab; VHL
MeSH Terms: conditions — von Hippel-Lindau Disease; Neoplasms; Macular Edema | interventions — Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab

SUMMARY:
This study will examine whether he drug ranibizumab can slow or stop the growth of angiomas (blood vessel tumors) in patients with Von Hippel-Lindau syndrome (VHL). Angiomas commonly develop in the back of the eye on the retina and the optic nerve in patients with VHL. Although these tumors are not cancerous, they may cause significant vision loss. Current treatments, including laser therapy, cryotherapy, and vitrectomy, may not be successful or possible for all patients. Ranibizumab decreases production of VEGF, a growth factor that is important for the formation of new blood vessels and that is elevated in patients with VHL. Preliminary findings from other studies suggest that ranibizumab can reduce retinal thickening caused by vessel and tumor growth and improve vision.

Patients 18 years of age and older with retinal angiomas due to VHL in one or both eyes and central vision loss of 20/40 or worse may be eligible for this study. Participants undergo the following tests and procedures:

* Medical history, physical examination, electrocardiogram (EKG) and blood tests.
* Eye examination, including eye pressure measurement and dilation of the pupils to examine the retina.
* Fluorescein angiography to evaluate the eye's blood vessels. For this test, a yellow dye is injected into an arm vein and travels to the blood vessels in the eyes. Pictures of the retina are taken using a camera that flashes a blue light into the eye. The pictures show if any dye has leaked from the vessels into the retina, indicating possible blood vessel abnormality.
* Optical coherence tomography to measure retinal thickness. The eyes are examined through a machine that produces cross-sectional pictures of the retina. These measures are repeated during the study to determine changes, if any, in retinal thickening.
* Stereoscopic color fundus photography to examine the back of the eye. The pupils are dilated with eye drops to examine and photograph the back of the eye.
* Electroretinogram (ERG) to measure electrical responses generated from within the retina. For this test, the patient sits in a dark room for 30 minutes with his or her eyes patched. Then, a small silver disk electrode is taped to the forehead, the eye patches are removed, the surface of the eye is numbed with eye drops, and contact lenses are placed on the eyes. The patient looks inside an open white globe that emits a series of light flashes for about 20 minutes. The contact lenses sense small electrical signals generated by the retina when the light flashes.
* Ranibizumab injections to treat ocular angiomas. Ranibizumab is injected through a needle into the eye's vitreous (gel-like substance that fills the inside of the eye). Seven injections are given over a 28-week period. Before each injection, the surface of the eye is numbed with anesthetic eye drops. This is followed by injection of another anesthetic into the lower portion of the eye in the clear tissue surrounding the white of the eye. After a few minutes, the ranibizumab is injected into the vitreous. Patients receive ranibizumab injections at the first visit (during enrollment) and again at 4, 8, 12, 16, 20 and 24 weeks after the first injection. At the 28-week visit, the doctor will determine if further treatment is needed. Patients can continue to have injections every 4 weeks until 1 year of follow-up (54 weeks).

At each injection visit, participants repeat most of the tests described above to evaluate the response to treatment and return a week later for another eye examination.

DETAILED DESCRIPTION:
Von Hippel-Lindau Syndrome (VHL) is an autosomal dominant heritable disorder in which multiple benign and malignant neoplasms and cysts of specific histopathologies develop in the kidney, adrenal gland, pancreas, brain, spinal cord, eye, inner ear, epididymis, and broad ligament. Retinal angioma may be one of the earliest manifestations of VHL disease and may lead to a significant decrease in visual acuity of the affected individual. These tumors rarely regress spontaneously. The main cause of vision loss is retinal edema, specifically macular edema secondary to enlargement of peripheral retinal angiomas or angiomas found on or around the optic disk. Treatment of retinal angiomas depends on the location and size of the lesions but typically consists of photocoagulation or cryotherapy. However, there is no proven effective therapy for the treatment of VHL ocular lesions on or surrounding the optic nerve or lesions in the peripheral retina too large to respond to the traditional therapies. The genetic mutation found in VHL disease up-regulates the production of vascular endothelial growth factor (VEGF). Immunochemical studies of the VHL ocular lesions, as well as others found elsewhere in the body show marked increase in VEGF. This open-label study will pilot the use of an anti-VEGF therapy, ranibizumab (rhuFab V2) in 5 participants to investigate the potential efficacy as a treatment for retinal angiomas associated with VHL. Participants will receive 7 intravitreal injections of study drug over a 6 month period, with the option of up to seven additional injections at the same dose and schedule during follow-up for a maximum period of 1 year after the initiation of treatment. The primary outcome will be a change in the best corrected visual acuity of 15 letters or more eight weeks after a participant receives the final study injection. The secondary outcomes will be a reduction in retinal thickening and leakage eight weeks after the participants receives the final study injection, and adverse events including local and systemic toxicities.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Participant must understand and sign the informed consent.
  2. Participant must be at least 18 years of age.
  3. Participant must have retinal angiomas secondary to VHL in one or both eyes.
  4. Participant must have either optic nerve tumors or peripheral tumors that have caused central vision loss of 20/40 or worse.
  5. Participant must have clear ocular media and adequate papillary dilation to permit good quality stereoscopic fundus photography.
  6. All women of childbearing potential must have a negative urine pregnancy test at baseline, and be willing to undergo urine pregnancy testing immediately prior to each injection, and monthly for at least 2 months following the last dose of ranibizumab.
  7. Women of child-bearing potential who are sexually active and men who are sexually active are required to use two forms of birth control during the course of the study.

EXCLUSION CRITERIA:

1. History (within past 5 years) or evidence of severe cardiac disease (apparent in electrocardiogram abnormalities, clinical history of unstable angina, acute coronary syndrome, myocardial infarction, revascularization procedure within 6 months prior to baseline, atrial or ventricular tachyarrythmias requiring ongoing treatment).
2. History of stroke within 12 months of study entry.
3. History within the past five years of a chronic ocular or periocular infection (including any history of ocular herpes zoster).
4. Current acute ocular or periocular infection.
5. Any major surgical procedure within one month of study entry.
6. Known serious allergies to fluorescein dye.
7. Previous participation in a clinical trial (for either eye) involving anti-angiogenic drugs (pegaptanib, ranibizumab, anecortave acetate, Protein Kinase C inhibitors, etc).
8. Previous intravitreal drug delivery (e.g., intravitreal corticosteroid injection or device implantation) in the study eye.
9. History of vitrectomy surgery in the study eye.
10. History of glaucoma filtering surgery in the study eye.
11. History of corneal transplant in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5
Dates: Start 2004-08-10; Study Completion 2007-08-15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Manski TJ, Heffner DK, Glenn GM, Patronas NJ, Pikus AT, Katz D, Lebovics R, Sledjeski K, Choyke PL, Zbar B, Linehan WM, Oldfield EH. Endolymphatic sac tumors. A source of morbid hearing loss in von Hippel-Lindau disease. JAMA. 1997 May 14;277(18):1461-6. doi: 10.1001/jama.277.18.1461. PMID 9145719